CLINICAL TRIAL: NCT07261358
Title: The Effect of Three-Dimensional Exercises ( Schroth Method ) on Trunk Muscle Endurance, Sleep Quality, and Quality of Life in Adolescents With Hyperkyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1024
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Spine Deformity; Kyphosis; Adolescent; Sleep Quality; Trunk Muscle Endurance
Keywords: postural kyphosis; sleep quality; trunk muscle endurance; adolescent spine deformity
MeSH Terms: conditions — Kyphosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-Dimensional Exercise Group (Experimental): Adolescents aged 12 to 18 years with a diagnosis of kyphosis will undergo a supervised three-dimensional exercise program based on the Schroth Method. The intervention is specifically tailored for adolescents with kyphosis and aims to improve postural alignment, increase spinal mobility, enhance back extensor muscle endurance, and restore trunk muscle balance. The program consists of 10 outpatient sessions (approximately 60 minutes each), delivered by a physiotherapist trained in the Schroth Method.
  Exercises include postural correction, rotational angular breathing techniques, stabilization strategies, and individualized corrective postures adapted to the patient's spinal deformity pattern. After completing the supervised sessions, participants will be instructed to continue performing the Schroth exercises as a home-based program for the remainder of the study period, with adherence monitored through exercise logs and outpatient follow-up.
  Interventions: Diagnostic Test: Kyphosis Study Form; Diagnostic Test: Scoliosis X-ray (Orthoroentgenogram); Diagnostic Test: Inclinometer Measurement; Diagnostic Test: Biering-Sorensen Test (Back Extensor Endurance Test)
- Control Group (Other): Adolescents aged 12 to 18 years with a diagnosis of kyphosis will be assigned to a home-based back extensor strengthening exercise program. Participants will receive detailed written and illustrated instructions on standardized back extensor strengthening exercises. After an initial instruction session, they will be asked to perform the exercises independently at home, every day per week, for the duration of the study period. Adherence will be monitored through exercise logs and outpatient follow-up visits.
  Interventions: Diagnostic Test: Kyphosis Study Form; Diagnostic Test: Scoliosis X-ray (Orthoroentgenogram); Diagnostic Test: Inclinometer Measurement; Diagnostic Test: Biering-Sorensen Test (Back Extensor Endurance Test)

INTERVENTIONS:
Diagnostic Test: Kyphosis Study Form — Kyphosis study form consisting of clinical and radiological measurements of patients aged 12-18 years who applied to the outpatient clinic with spine deformity will be filled in detail.
Diagnostic Test: Scoliosis X-ray (Orthoroentgenogram) — Adolescents aged 12-18 years presenting to the scoliosis outpatient clinic will undergo a standardized physical examination. Posture will be assessed in standing position from both anterior and lateral views in front of a posture chart. In patients where thoracic kyphosis is clinically suspected, a standing orthoroentgenogram (whole-spine radiograph) will be requested. On these radiographs, thoracic kyphosis angles will be measured to confirm the diagnosis and establish baseline values. Clinical and radiological data will be recorded in detail before study group allocation.
Diagnostic Test: Inclinometer Measurement — Thoracic kyphosis angle will also be assessed using a bubble inclinometer during physical examination. The participant will stand in a relaxed upright position, and the inclinometer will be placed over the spinous processes from T3 to T12 to measure the sagittal alignment of the thoracic spine. Three consecutive measurements will be taken for each participant, and the mean value will be recorded for analysis. This provides a reliable clinical estimate of thoracic kyphosis in addition to radiographic assessment.
Diagnostic Test: Biering-Sorensen Test (Back Extensor Endurance Test) — The Biering-Sorensen test is a standardized clinical assessment used to evaluate the isometric endurance of the trunk extensor muscles. During the test, the participant lies prone on an examination table with the upper edge of the iliac crests aligned with the edge of the table. The lower body (pelvis, knees, and ankles) is stabilized using straps or manual fixation. The upper body is extended horizontally beyond the edge of the table, with the arms crossed over the chest. The participant is instructed to maintain the unsupported horizontal trunk position for as long as possible without assistance.
  The outcome is recorded as the duration, in seconds, that the participant can hold the trunk in a straight horizontal alignment before fatigue, deviation from the position, or voluntary termination occurs.

SUMMARY:
Adolescence is a critical period for spinal growth, and progression of thoracic hyperkyphosis may lead to pain, weak trunk muscles, sleep disturbances, and reduced quality of life. This study aims to investigate the effects of three-dimensional exercise program based on the Schroth Method on trunk muscle endurance, thoracic kyphosis angle, pain, sleep quality and quality of life in adolescents aged 12-18 years with hyperkyphosis.

DETAILED DESCRIPTION:
Childhood and adolescence are critical developmental stages characterized by rapid spinal growth, as well as the formation of postural habits and the musculoskeletal system. During this process, various spinal deformities may arise due to neuromuscular, structural, postural, or functional causes, and if not addressed in a timely manner, they can lead to permanent postural abnormalities carried into adulthood.

Thoracic kyphosis is the physiologically present forward curvature of the spine in the sagittal plane and is generally considered normal within the range of 20°-45°. However, when this angle exceeds 45°, it is referred to as hyperkyphosis. Hyperkyphosis can develop due to many different causes, such as postural abnormalities, muscle imbalances, and vertebral developmental anomalies. This deformity can become more pronounced, especially during adolescence when growth spurts occur.

The progression of hyperkyphosis that emerges during the developmental period can lead to serious clinical consequences in children and adolescents, including aesthetic concerns, weak trunk muscles, pain around the spine, sleep disorders, and a decline in quality of life. Timely diagnosis and effective rehabilitation of adolescent hyperkyphosis are critical in controlling the progression of the deformity and preventing functional loss.

The literature reports that exercise-based approaches are effective in treating kyphosis in this age group. Schroth exercises, in particular, are a specialized physical therapy protocol used in the treatment of 3-dimensional scoliosis and kyphosis. They offer individualized, breathing-integrated postural correction techniques that target interplanar asymmetry of the spine. With this approach, patients are taught positioning to actively correct spinal segments, proprioceptive awareness, and breathing control. The Schroth method aims not only at passive posture correction but also at reestablishing muscle balance and maintaining correct posture in daily life.

In this context, Schroth exercises, which specifically target 3-dimensional spinal correction, are among the interventions frequently recommended in the literature.

The aim of this study is to evaluate the effect of Schroth exercises on back muscle endurance, thoracic kyphosis angle, pain, quality of life, and sleep in adolescents with hyperkyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 and 18 years of age
* Presence of thoracic kyphosis with a T3-T12 Cobb angle ≥45° measured on a lateral thoracic radiograph
* Sufficient physical and cognitive ability to actively participate in the exercise protocol for at least 3 months
* Adequate communication and cognitive capacity to understand the educational materials provided
* Ability and willingness to regularly complete the exercise log throughout the study period

Exclusion Criteria:

* Scoliosis with a Cobb angle >10° in the coronal plane
* Presence of structural spinal deformities such as vertebral fracture, spondylolisthesis
* History of previous spinal surgery
* Neuromuscular disorders that may affect the spine (e.g., cerebral palsy, muscular dystrophy)
* Structural or functional pathologies involving the spine, pelvic complex, or shoulder girdle
* Balance disorders such as vestibular dysfunction, vertigo, or other conditions affecting postural control
* Inability to comply with the exercise protocol due to intellectual disability, severe behavioral disorders, or significant communication impairments
* Participation in professional-level sports activities that may influence exercise capacity or musculoskeletal function
* Presence of serious cardiopulmonary diseases (e.g., congenital heart disease, pulmonary hypertension)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Biering-Sorensen Test (Back Extensor Endurance Test) | Assessments will be performed at baseline (one day before the exercise program ), at 1 month and at 3 months after the initiation of exercises.
  The Biering-Sorensen test is a standardized clinical assessment used to evaluate the isometric endurance of the trunk extensor muscles. During the test, the participant lies prone on an examination table with the upper edge of the iliac crests aligned with the edge of the table. The lower body (pelvis, knees, and ankles) is stabilized using straps or manual fixation. The upper body is extended horizontally beyond the edge of the table, with the arms crossed over the chest. The participant is instructed to maintain the unsupported horizontal trunk position for as long as possible without assistance. The outcome is recorded as the duration, in seconds, that the participant can hold the trunk in a straight horizontal alignment before fatigue, deviation from the position, or voluntary termination occurs.
Thoracic Kyphosis Angle (Inclinometer Measurement) | Assessments will be performed at baseline (one day before the exercise program), at 1 month and at 3 months after the initiation of exercises.
  Thoracic sagittal alignment will be assessed using a bubble inclinometer placed over the spinous processes from T3 to T12 while the participant stands in a relaxed upright position. Three consecutive measurements will be performed for each participant, and the mean value will be recorded for analysis. This clinical method provides a reliable and non-invasive estimate of thoracic kyphosis angle in adolescents.

SECONDARY OUTCOMES:
Thoracic Kyphosis Angle (Inclinometer Measurement) | Assessments will be performed at baseline (one day before the exercise program), at 1 month and at 3 months after the initiation of exercises.
  Thoracic sagittal alignment will be assessed using a bubble inclinometer placed over the spinous processes from T3 to T12 while the participant stands in a relaxed upright position. Three consecutive measurements will be performed for each participant, and the mean value will be recorded for analysis. This clinical method provides a reliable and non-invasive estimate of thoracic kyphosis angle in adolescents.
Pittsburgh Sleep Quality Index (PSQI) | Assessments will be performed at baseline (one day before the exercise programme ), at 1 month and at 3 months after the initiation of exercises.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-reported questionnaire that evaluates sleep quality and disturbances over the previous month. The PSQI consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored on a scale of 0 to 3, yielding a total score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Adolescent Insomnia Questionnaire (AIQ) | Assessments will be performed at baseline (one day before the exercise programme ), at 1 month and at 3 months after the initiation of exercises.
  Insomnia symptoms will be assessed using the Adolescent Insomnia Questionnaire (AIQ), a validated self-reported instrument specifically developed for adolescents to evaluate insomnia severity and sleep difficulties. The AIQ consists of 13 items covering three main domains: difficulties initiating sleep, difficulties maintaining sleep, and early morning awakenings. Each item is rated on a 0-4 Likert scale, with higher scores indicating greater severity of insomnia symptoms. The AIQ has been shown to be reliable and valid for assessing insomnia in adolescents.
Visual Analog Scale | Assessments will be performed at baseline (one day before the exercise programme ), at 1 month and at 3 months after the initiation of exercises.
  Pain intensity will be assessed using the Visual Analog Scale (VAS) with facial expression illustrations. This tool consists of a series of facial expressions ranging from a smiling face indicating "no pain" (score 0) to a crying face indicating "worst pain" (score 10). Participants will be asked to select the face that best represents their current level of back pain. Scores will be recorded on a 0-10 scale, with higher scores reflecting greater pain severity.
Scoliosis Research Society-22 Questionnaire | Assessments will be performed at baseline (one day before the exercise programme ), at 1 month and at 3 months after the initiation of exercises.
  Health-related quality of life will be evaluated using the Scoliosis Research Society-22 (SRS-22) Questionnaire. The SRS-22 is a validated patient-reported outcome measure that consists of 22 items grouped into five domains: Function/Activity, Pain, Self-image/Appearance, Mental Health, and Satisfaction with Management. Each item is scored on a 5-point Likert scale, where higher scores indicate better health status and quality of life. Domain scores and the total score will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yılmaz Yalçınkaya, MD,Professor, Study Director — Gaziosmanpaşa Training and Research Hospital Physical Rehabilitation Department
Locations (1):
- Gazisomanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schreiber S, Parent EC, Moez EK, Hedden DM, Hill D, Moreau MJ, Lou E, Watkins EM, Southon SC. The effect of Schroth exercises added to the standard of care on the quality of life and muscle endurance in adolescents with idiopathic scoliosis-an assessor and statistician blinded randomized controlled trial: "SOSORT 2015 Award Winner". Scoliosis. 2015 Sep 18;10:24. doi: 10.1186/s13013-015-0048-5. eCollection 2015. PMID 26413145